CLINICAL TRIAL: NCT01299818
Title: Assessment of Central Pain in Patients Who Undergo Spinal Surgery and Influence in Surgery Outcome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Jacob Ablin, TASMC
Other Study IDs: 0104-10-TLV
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Spinal Surgery; Pain
Keywords: central pain; spine surgey; outcome; patients undergo spinal surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- spinal surgery: patients who undergo spinal surgery

SUMMARY:
* Pain is one of the most common concerns for which patients seek medical attention.
* Pain is usually understood as symptom that reflects peripheral organic damage. Many patients experience pain, often chronically, independently of any underlying cause such as chronic regional pain syndromes (irritable bowel syndrome, temporo-mandibular pain syndrome, chronic headache or chronic low back pain)or diffuse like in fibromyalgia. In all those "functional" syndromes, accumulated evidence supports involvement of central pain processing systems, hypothalamic pituitary adrenal axes and autonomic nervous system, and are now referred as central pain conditions.
* Other patients suffers from chronic pain caused by damage or inflammation in peripheral tissues, but also experienced more diffuse pain, not directly explained by peripheral damage, that further aggravates pain and function. This is illustrated by the high prevalence of fibromyalgia observed in patients with rheumatoid arthritis, osteoarthritis or ankylosing spondylitis for example.

These pain conditions are now understood as combinations of peripheral, neuropathic and central pain.

The investigators aimed to focus in this study in patients that are candidates to spinal surgery and suffer from low back pain and/or radiculopathy. Pain in these patients may arise from damage to nerves - neuropathic pain- , to musculoskeletal structures - peripheral pain-, and may also reflects alteration in central pain processes.

In these patients, spine surgery is usually performed to improve quality of life, decrease pain and avoid neurological deficits. Evaluation of surgical outcome includes objective measures such as neurological findings and radiographic evaluation, and subjective measures including patient self-assessments for pain and quality of life and psychological changes.

The aim of this study is to evaluate patients who undergo spinal surgery for presence of central pain and central sensitization symptoms and evaluate their influence on these surgical outcomes

ELIGIBILITY:
Inclusion Criteria:

* candidates to spinal surgery attending the spine clinic
* able to give inform consent

Exclusion Criteria:

* pregnant women
* children under 18
* current infection in spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients sufferring of cervicalgia and/or low back pain and/or radiculopathy that are candidates to spinal surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
evaluation of surgery outcome including pain and functionnal ability | 3 months
  evaluation of course of surgery, use of analgesics medications, report of pain intensity, length of hospital stay, questionnaires of health status and functionnal index, physical examination and dolorimetric evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Ablin, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Ablin K, Clauw DJ. From fibrositis to functional somatic syndromes to a bell-shaped curve of pain and sensory sensitivity: evolution of a clinical construct. Rheum Dis Clin North Am. 2009 May;35(2):233-51. doi: 10.1016/j.rdc.2009.06.006. PMID 19647139